CLINICAL TRIAL: NCT02767141
Title: Understanding the Interdependencies Among Three Types of Coping Strategies Used by Very Low Food Security Households With Children
Brief Title: Coping Strategies Used by Food Insecure Households
Status: Completed | Type: Observational
Sponsor: RTI International (Other)
Responsible Party: Sponsor
Other Study IDs: 13224
Record Dates: First submitted 2016-04-11; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Food Insecurity
Keywords: Hunger; food insecurity; behaviors
MeSH Terms: conditions — Behavior | interventions — Coping Skills

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Coping Strategies — Coping strategies for households in the US with food insecurity

SUMMARY:
Children without consistent access to sufficient and nutritious food show sustained disadvantages. To improve food security, households utilize three types of coping strategies- participating in governmental feeding and financial assistance programs; obtaining food from nongovernment providers; and using individually developed strategies. To understand the interdependencies among strategies and decision-making processes used to select them, the investigators conducted a two-phased, mixed-methods study using a socio-ecological theoretical framework. First, employing a cross sectional, observational design the investigators administered in-person surveys to 320 adults in very low food secure (VLFS) households with children. Over 1 year later, the investigators repeated select questions and conducted in depth interviews with a cohort (n=28) of participants. Descriptive statistics defined magnitude of associations among strategies. Following bivariate analysis, the investigators assessed interdependencies and factors affecting relationships with log-linear models. The investigators analyzed interviews using an hierarchically ordered, analytical coding structure. With Qualitative Comparative Analysis (QCA), the investigators developed typologies of VLFS and created models treating food security as an outcome. The association of soup kitchen use and nutritionally risky behavior was altered by Supplemental Security Income (SSI) or Social Security Disability Insurance (SSDI). Food safety-related risky behavior level related to intensity of food pantry use by participation in school food programs. Supplemental Nutrition Assistance Program (SNAP) did not affect the association between soup kitchen use and risky food safety behaviors. Key interview constructs included becoming and being short of food; coping strategies; decisions used to inform choice of strategies; and managing a devalued social status. Improved income stability was a necessary condition for improving food security.

DETAILED DESCRIPTION:
Food insecurity is a serious issue facing households in the United States. In 2012, the time this study was begun, the U.S. Department of Agriculture reported that almost 15% of U.S. households and one in five households with children were considered to be food insecure. Over one third of these experienced very low food security (VLFS), with multiple indicators of disrupted eating patterns due to inadequate resources. These statistics are of particular concern because children without consistent access to sufficient and nutritious food show sustained disadvantages, including effects on cognition, academic performance, long-term nutritional status, and psychosocial development. To improve their food security, households utilize three types of coping strategies- (1) participating in federal feeding and financial assistance programs ("safety net"), (2) obtaining food from nongovernment Emergency Food Providers (EFPs), and (3) using individually developed coping strategies. The objectives of this study related to developing a better understanding of the coping strategies that VLFS households with children use to ensure that their households have sufficient food. Specifically, the study addressed two main research questions: What are the interdependencies among three types of coping strategies: participating in federal feeding and financial assistance programs ("safety net"), obtaining food from EFPs, and using individually developed coping strategies. What decision-making processes do people in VLFS households with children use when selecting coping strategies to ensure that their households have sufficient food? The investigators conducted a two-phased mixed-methods study of coping strategies used by VLFS households with children <18 years in North Carolina (NC), using a socio-ecological theoretical framework to guide their hypotheses, methods, and analyses. For phase I, the investigators employed a cross sectional, observational design. The investigators used a two-stage sample to recruit 320 clients of service providers who offer assistance to people with limited resources within eight NC counties with the highest food insecurity rates. Trained interviewers administered in-person a survey interview asking clients socio-demographic questions and about their use of three categories of coping strategies. Using a longitudinal design, more than a year after Phase I, in Phase II, the investigators completed in depth interviews with a cohort (n=28) of Phase I participants, selected using maximum variation sampling. During the largely unscripted interviews, participants were asked a select number of close ended questions from Phase I, including the 18 item food security module, to assess changes over the past year and permit comparisons between times one and two. To address the first question, two by two and multi-dimensional contingency tables were constructed to analyze the interdependencies among the three types of coping strategy outcomes. Descriptive statistics (odds ratios, counts and percentages) were performed to define the magnitude of the association among coping strategies. Fisher's exact tests and Chi-square statistics were then employed to assess the statistical significance of the interdependency among the outcomes. To further determine the interdependencies among the three coping strategies, and to assess how individual and household-level factors affect those interdependencies, the investigators employed log-linear models. To address the second research question, the investigators formulated a hierarchically ordered, analytical coding structure that reflected key decision-making constructs (e.g., knowledge of coping strategies, perception of risk of accessibility and availability of coping strategies, barriers to participation in "safety net" programs) and examined the results in terms of the key constructs. Lastly, responses to both sets of questions were jointly reviewed using Qualitative Comparative Analysis (QCA), a mixed-methods analysis technique. The investigators implemented a conventional, crisp set for (1) developing typologies of households and individuals experiencing very low food insecurity, and (2) exploring pathways to improving food security status among participants in the follow-up interviews. All procedures involving human participants was reviewed and approved by RTI International's Institutional Review Board (IRB).

ELIGIBILITY:
Inclusion Criteria::

* 18 years of age or older
* responsible for getting food for household
* household assessed to have very low food security
* children <18 in household
* consent to participate

Exclusion Criteria:

* less than 18 years of age
* never responsible for getting food for household
* no children <18 in household
* do not consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 320 clients of service providers who offer assistance to people with limited resources within eight North Carolina counties with the highest food insecurity rates. Using a longitudinal design, more than a year after Phase I, in Phase II, the investigators completed in depth interviews with a cohort (n=28) of Phase I participants
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Identify participants who have used at least one target coping strategy | Initial contact
  Participants were administered a survey to document their use of at least one target coping strategy within the last twelve months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Anater, Ph.D., Principal Investigator — RTI International
Locations (26):
- United States (26):
  - Christians United Outreach Center, Asheboro, North Carolina
  - Salvation Army, Asheboro, North Carolina
  - Bladen Family Support, Clarkton, North Carolina
  - Bladen Crisis Assistance Center, Elizabethtown, North Carolina
  - Liberty Baptist, Ellenboro, North Carolina
  - Chase Corner UMC Ministries, Forest City, North Carolina
  - Grace Country Kitchen at Grace of God Rescue Mission, Forest City, North Carolina
  - St. John's UMC, Gibson, North Carolina
  - Higher Dimensions, Laurel Hill, North Carolina
  - Church Community Service of Scotland County, Laurinburg, North Carolina
  - Laurinburg Hope In Christ Ministries, Laurinburg, North Carolina
  - Robeson County Church and Community Center, Lumberton, North Carolina
  - Living Bread Holiness Church, New Bern, North Carolina
  - Religious Community Services, New Bern, North Carolina
  - Sacred Pathways, Pembroke, North Carolina
  - Little White Country Church, Rutherfordton, North Carolina
  - New Bethel Church, Saint Pauls, North Carolina
  - Black Swamp Church of Christ, Williamston, North Carolina
  - Holy Trinity Church, Williamston, North Carolina
  - Liberty Christian Center Food Pantry, Williamston, North Carolina
  - Unlimited Care, Williamston, North Carolina
  - Christ Deliverance Tabernacle Ministries, Wilson, North Carolina
  - New Christian Food Pantry, Wilson, North Carolina
  - Salvation Army, Wilson, North Carolina
  - Wilson County Interfaith Services: Hope Station, Wilson, North Carolina
  - Willson Praise & Worship Church, Wilson, North Carolina